CLINICAL TRIAL: NCT02878980
Title: An Exercise Intervention Trial to Reduce Symptoms & Improve Clinical Outcomes of Platinum-Based Treatment in Ovarian Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility issues
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15388; NCI-2016-01183 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15388 (Other: City of Hope Medical Center)
Record Dates: First submitted 2016-08-02; First posted 2016-08-25 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (exercise intervention) (Experimental): Patients undergo supervised 1-on-1 exercise sessions for 60 minutes on day 1.Treatment repeats every 3 weeks for up to 18 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive a home-based exercise prescription including instructions for keeping patients' heart rate within 50-80% maximum.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo supervised 1-on-1 exercise sessions
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well an exercise intervention works in reducing symptoms and improving clinical outcomes in patients with ovarian cancer undergoing platinum-based chemotherapy. Exercise may "train" the body to repair deoxyribonucleic acid (DNA) damage more efficiently, which may reduce symptoms related to platinum-based chemotherapy, improve quality of life, increase survival, and decrease recurrence rates in patients with ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of recruiting and enrolling newly diagnosed epithelial ovarian cancer patients who have undergone debulking surgery and will be starting platinum-based chemotherapy, to an exercise trial.

II. To evaluate adherence to the data collection and exercise trial protocol. It is necessary to determine the feasibility of collecting tablet-based questionnaire data and blood samples at multiple time points in one visit. It is also critical to determine whether the exercise intervention is feasible in this patient population.

SECONDARY OBJECTIVES:

I. To examine changes in DNA repair function before and after a single exercise session.

II. To examine changes in DNA repair function, body composition, quality of life, symptoms and patient satisfaction with care over the treatment time course.

III. To examine the effect of the exercise intervention on these measurements.

IV. To follow the patients an additional 12-months for clinical outcomes defined as death, cancer recurrence, or new primary cancer.

OUTLINE: Patients undergo supervised 1-on-1 exercise sessions for 60 minutes on day 1.Treatment repeats every 3 weeks for up to 18 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive a home-based exercise prescription including instructions for keeping patients' heart rate within 50-80% maximum.

After completion of study, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Women who have been newly diagnosed with a first primary, epithelial ovarian cancer, have undergone surgical debulking and who will be treatment according to the Armstrong method
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately.
* Newly diagnosed, primary, epithelial ovarian cancer
* Have undergone surgical debulking
* Will be treated according to the Armstrong method
* Read and understand English
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to the data collection and exercise trial protocol, defined as the number of sessions attended, questionnaires completed, and blood samples completed | 18 weeks
Feasibility of recruiting and enrolling patients to an exercise trial, defined as the number of people contacted, eligible consented and enrolled | 12 months

SECONDARY OUTCOMES:
Change in body composition | Baseline to 18 weeks
  Will be analyzed using paired t-tests. Data from women in course 1 will be compared to data in women in course 6.
Change in DNA repair function, assessed by host reactivation assays | Before single exercise session to after single exercise session, assessed up to 12 months
  Will be analyzed using paired t-tests
Change in DNA repair function, assessed by host reactivation assays | Baseline to 18 weeks
  Will be analyzed using paired t-tests. Data from women in course 1 will be compared to data in women in course 6.
Change in quality of life, assessed by questionnaires | Baseline to 18 weeks
  Will be analyzed using paired t-tests. Data from women in course 1 will be compared to data in women in course 6.
Change in symptoms, assessed by National Comprehensive Cancer Network Functional Assessment of Cancer Therapy Ovarian Symptom Index-18 version 2 | Baseline to 18 weeks
  Will be analyzed using paired t-tests. Data from women in course 1 will be compared to data in women in course 6.
Change in treatment satisfaction, assessed by Functional Assessment of Chronic Illness Therapy-Treatment Satisfaction-General | Baseline to 18 weeks
  Will be analyzed using paired t-tests. Data from women in course 1 will be compared to data in women in course 6.
Clinical outcome follow-up defined as death, cancer recurrence, or new primary cancer | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Clague DeHart, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States